CLINICAL TRIAL: NCT05590637
Title: A Pragmatic Randomized Trial Comparing Antipsychotics in Lewy Body Disease
Brief Title: Comparing Antipsychotic Medications in LBD Over Time
Acronym: CAMELOT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-0198H
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease Psychosis; Dementia With Lewy Bodies
Keywords: quetiapine; pimavanserin; psychosis; hallucinations; delusions
MeSH Terms: conditions — Lewy Body Disease; Psychotic Disorders; Hallucinations; Delusions | interventions — pimavanserin; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- quetiapine (Active Comparator): Elderly patients with dementia-related psychosis will be treated with quetiapine, an atypical antipsychotic indicated for the treeatment of: schizophrenia, bipolar I manic episodes and bipolar depressive episodes.
  Interventions: Drug: Quetiapine
- pimavanserin (Active Comparator): Elderly patients with dementia-related psychosis will be treated with pimavanserin, an atypical antipsychotic indicated for treatment of hallucinations and delusions associated with Parkinson's disease.
  Interventions: Drug: Pimavanserin

INTERVENTIONS:
Drug: Pimavanserin — Dosage choice and further medication management will be at the discretion of the treating clinician, per routine clinical practice.
  Other Names: Nuplazid
  Arms: pimavanserin
Drug: Quetiapine — Dosage choice and further medication management will be at the discretion of the treating clinician, per routine clinical practice.
  Other Names: Seroquel
  Arms: quetiapine

SUMMARY:
The primary objective of this study is to determine whether treatment with pimavanserin or quetiapine is associated with a greater improvement in psychosis when used in a routine clinical setting to treat hallucinations and/or delusions due to Parkinson's disease (PD) or dementia with Lewy bodies (DLB) - collectively referred to as Lewy body disease (LBD).

DETAILED DESCRIPTION:
Psychosis (hallucinations and delusions) is a common problem in Parkinson's disease (PD) and dementia with Lewy bodies (DLB). PD is a common neurodegenerative disorder that causes movement, cognitive, and psychiatric symptoms. DLB is a similar disorder, though causes more severe cognitive and psychiatric problems. Psychosis is highly prevalent among people with PD and DLB, often manifesting as visual hallucinations or paranoid delusions. Up to 60% of people with PD will experience psychosis over the course of their disease. Psychosis is associated with increased mortality, caregiver burden, and poorer quality of life.

More study is needed to determine the best way to treat psychosis in PD and DLB. Currently, both quetiapine and pimavanserin are used in clinical practice for psychosis in PD and DLB. However, few comparison studies have been done and it is unclear if one medication is superior to the other. This will be a clinical trial comparing quetiapine and pimavanserin among patients with psychosis due to PD or DLB requiring initiation of a medication. Patients will be randomized to quetiapine or pimavanserin and improvement in psychosis at 6 months will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the neurology clinic at UT Health San Antonio
* Diagnosed with psychosis due to PD or DLB
* Requiring initiation of an antipsychotic medication
* Clinical equipoise between quetiapine and pimavanserin must exist
* The prescribing provider must be comfortable prescribing and managing both quetiapine and pimavanserin

Exclusion Criteria:

* Medical contraindication to either medication
* Caregiver unavailable to complete NPI-Q
* Currently taking an antipsychotic medication
* Prescribing provider unwilling to manage either medication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatry Inventory Questionnaire (NPI-Q), Hallucinations + Delusions (H+D) | Baseline to 6 months
  Change in the Hallucinations + Delusions sub-score of the neuropsychiatric inventory questionnaire. Each NPI-Q item is scored by severity (1-3), and distress to caregiver (0-5), then added together (range 0-8) with a higher score indicating greater severity.

SECONDARY OUTCOMES:
Neuropsychiatry Inventory Questionnaire (NPI-Q) total score | Baseline to 6 months
  Change in the total neuropsychiatric inventory questionnaire score, which includes 12 items, each scored from 0-8 with a higher score indicating more severe symptoms.
Neuropsychiatry Inventory Questionnaire (NPI-Q) (anxiety) | Baseline to 6 months
  Change in the neuropsychiatric inventory questionnaire item for anxiety, scored from 0-8 with a higher score indicating more severe anxiety.
Neuropsychiatry Inventory Questionnaire (NPI-Q) (agitation) | Baseline to 6 months
  Change in the neuropsychiatric inventory questionnaire for agitation, scored from 0-8 with a higher score indicating more severe agitation.
Neuropsychiatry Inventory Questionnaire (NPI-Q) (nighttime behaviors) | Baseline to 6 months
  Change in the neuropsychiatric inventory questionnaire for sleep disturbance, scored from 0-8 with a higher score indicating more severe sleep disturbances.
Mortality | 6 months
  Number of subjects who survived until the 6 month study assessment visit
Time to discontinuation of per-protocol medication | Baseline to 6 months
  Will examine whether participants continued the chosen medication until study completion or if they either discontinued the study medication or added the other study medication.
MDS-UPDRS part 3 | Baseline to 6 months
  Unified Parkinson's Disease Rating Scale, motor score. The motor examination scale consists of 33 items graded 0-4 points with an overall possible score of 0-132 points. A higher score indicates a higher burden of motor symptoms.
CGIC, PGIC, CGI-C:CVR | Baseline to 6 months
  Clinician, patient, and caregiver global impressions of change. Each is a single item assessment rated from 1 (very much improved) to 7 (very much worse). A higher score indicates worsening symptoms.

OTHER OUTCOMES:
Medication out-of-pocket cost | Baseline to 6 months
  Amount of out of pocket costs spent on medications during the study
NPI-Q caregiver portion | Baseline to 6 months
  Change in the total of the caregiver distress items of the neuropsychiatric inventory. The scale contains 12 items, each scored from 0-5 (least to most distress). Possible scores Range from 0-60 with a lower score indicating less caregiver distress
Patient contact | Baseline to 6 months
  Number of between visit patient encounters (phone, EMR messages)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Horn, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (2):
- United States (2):
  - University Health System, San Antonio, Texas
  - UT Health Science Center - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran N, Wang CP, Seshadri S, Coss P, Vaou OE, Saadatpour L, Paiz C, Solis D, Grimaldo J, Erskine S, Horn S. Pragmatic trial design enhances diversity and retention among research participants with Lewy body diseases. NPJ Dement. 2026;2(1):10. doi: 10.1038/s44400-026-00059-x. Epub 2026 Feb 2. PMID 41640857